CLINICAL TRIAL: NCT01210872
Title: Impact of Quality of Life Assessment in Routine Oncology Practice for Head and Neck's Cancer Patients, Treated by Radiotherapy: Impact on the Satisfaction With Care, the Health Related Quality of Life and on the Toxicity
Brief Title: Quality-Of-Life Assessment in Patients With Head and Neck Cancer Treated With Radiation Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CGFL-QDV; CDR0000683850 (Registry Identifier: PDQ (Physician Data Query)); CGFL-AFSSAPS-2008-A01468-47; EU-21061
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2010-09

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage I lymphoepithelioma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III verrucous carcinoma of the larynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms

INTERVENTIONS:
Other: questionnaire administration
Procedure: quality-of-life assessment
Procedure: standard follow-up care

SUMMARY:
RATIONALE: Gathering information over time about patients' quality-of-life and satisfaction with care may help doctors plan the best treatment and help patients live more comfortably.

PURPOSE: This randomized clinical trial is studying quality-of-life assessment in patients with head and neck cancer treated with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the impact of quality-of-life assessment in routine oncology practice on satisfaction with care, health-related quality-of-life, and toxicity in patients with primary nonmetastatic head and neck cancer treated with radiotherapy.

Secondary

* To evaluate the feasibility of using quality-of-life tools in routine oncology practice.
* To evaluate the impact on the occurrence of toxicity.
* To determine the impact on overall survival.
* To study the concordance between the toxicity reported by the clinician and those reported by the patient quality-of-life questionnaires.

OUTLINE: Patients are stratified according to sex, tumor localization, and TNM stage. Patients are randomized to 1 of 2 arms.

* Arm I: Patients complete quality-of-life questionnaires (EORTC tools only, including EORTC QLQ-SAT32, EORTC QLQ-C30, and specific module QLQ-H&N35/Euroqol EQ-5D) before each consultation with the clinician for one year.
* Arm II: Patients undergo standard follow-up care comprising consultation with the clinician for one year.

After completion of study, patients are followed up every 3 months for 1 year and then at 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary nonmetastatic head and neck cancer
* No other primary cancer localizations
* No second tumor localization at the time of diagnosis
* Must be planning to be treated initially with radiotherapy

PATIENT CHARACTERISTICS:

* No cognitive impairment or psychiatric history
* No history of other cancer

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of care (EORTC QLQ-SAT32)
Quality of life (EORTC QLQ-C30 and specific module QLQ-H&N35/Euroqol EQ-5D)

SECONDARY OUTCOMES:
Toxicity (occurrence and length) according to NCI-CTC version 3.0
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Maingon, MD, Study Chair — Centre Georges Francois Leclerc; Franck Bonnetain, PhD — Centre Georges Francois Leclerc
Locations (1):
- Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon, France